CLINICAL TRIAL: NCT04989816
Title: A Single-arm Study of Trastuzumab Deruxtecan (T-DXd) Monotherapy for Patients With HER2-expressing Locally Advanced or Metastatic Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma Who Have Received 2 or More Prior Regimens (DESTINY-Gastric06)
Brief Title: Study of T-DXd Monotherapy in Patients With HER2-expressing Locally Advanced or Metastatic Gastric or GEJ Adenocarcinoma Who Have Received 2 or More Prior Regimens
Acronym: DG-06
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9676C00002
Record Dates: First submitted 2021-07-14; First posted 2021-08-04 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma
Keywords: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma; HER2; Trastuzumab; Deruxtecan; T-DXd; DS-8201a; ERBB2
MeSH Terms: conditions — Adenocarcinoma; Stomach Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T-DXd arm (Experimental): T-DXd monotherapy
  Interventions: Drug: Trastuzumab Deruxtecan

INTERVENTIONS:
Drug: Trastuzumab Deruxtecan — Trastuzumab deruxtecan (T-DXd) by intravenous infusion
  Other Names: DS8201a; AZD4552; T-DXd

SUMMARY:
This is a Phase II, open-label, single-arm, multicentre, study in China assessing the efficacy and safety of T-DXd in participants with HER2-expressing advanced gastric or GEJ adenocarcinoma who have received at least 2 prior regimens including a fluoropyrimidine agent and a platinum agent

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age
2. Pathologically documented gastric or GEJ adenocarcinoma
3. Disease progression on or after ≥ 2 prior platinum and fluoropyrimidine agents for advanced/metastatic disease
4. ECOG PS 0-1
5. Willing and able to provide an adequate newly-acquired tumour sample for confirmation of HER2 status
6. LVEF ≥ 50%

Exclusion Criteria:

1. Pleural effusion, ascites or pericardial effusion that requires drainage, peritoneal shunt, or Cell-free and CART. Drainage and CART.
2. Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring steroids
3. Active primary immunodeficiency, known HIV, active HBV, HCV infection.
4. Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals.
5. History of non-infectious pneumonitis/ILD, current ILD, or where suspected ILD that cannot be ruled out by imaging at screening.
6. Lung-specific intercurrent clinically significant severe illnesses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Lanzhou
  - Research Site, Nanchang
  - Research Site, Nanchong
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Suzhou
  - Research Site, Wuhan
  - Research Site, Xiamen
  - Research Site, Yinchuan
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . A Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9676C00002&attachmentIdentifier=2daaaa16-936a-4e55-b281-20c4d5121fc3&fileName=d9676c00002-csp-v2__Redacted_BX_ZQ_27May24_(1).pdf&versionIdentifier=
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9676C00002&attachmentIdentifier=8753c80f-24f8-440e-97aa-cfa37faf5223&fileName=d9676c00002-sap-ed-4_Redacted_12Jun24.pdf&versionIdentifier=
- See also: CSR Synopsis redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9676C00002&attachmentIdentifier=ad306a1d-acf7-433e-bbdf-fe2676eb9672&fileName=d9676c00002-clinical-study-report-Synopsis-Redacted-12Jun24.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T-DXd Arm
Started (Enrolled) | 95
Received Treatment | 95
Completed | 15
Not Completed | 80
Not completed — Death | 77
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 95
Age, Continuous [Median (Full Range); unit: Years] | 60 [28 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 95
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 95
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate by RECIST 1.1 Based on Independent Central Review (ICR)
Description: Confirmed ORR is defined as the proportion of participants who have a confirmed CR or confirmed PR, as determined by ICR per RECIST 1.1.
Time Frame: Tumour assessments every 6 weeks from 1st dose of treatment until Recist 1.1 defined radiological progressive disease. Assessed up to a maximum of 19.3 months
Population: HER2-positive Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 73
Percentage of Participants | 28.8 [18.8 to 40.6]

2. Primary Outcome: Best Objective Response Rate by RECIST 1.1 Based on Independent Central Review (ICR)
Description: The best response based on the overall visit responses from each RECIST 1.1 assessment or the last evaluable assessment in the absence of RECIST 1.1 progression
Time Frame: as for outcome 1
Population: HER2-positive Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 73
Participants
  Complete response (confirmed after at least 4 weeks) | 1
  Partial response (confirmed after at least 4 weeks) | 20
  Stable disease | 37
  Progression | 14
  Not evaluable | 1

3. Secondary Outcome: Progression-free Survival (PFS) Based on Independent Central Review (ICR)
Description: PFS based on ICR is defined as the time from date of enrolment until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdraws from therapy or receives another anti-cancer therapy prior to progression
Time Frame: Tumour assessments every 6 weeks from 1st dose of treatment until Recist 1.1 defined radiological progressive disease. Assessed up to a maximum of 22 months
Population: HER2-positive Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 73
Months | 5.7 [4.0 to 6.8]

4. Secondary Outcome: Progression-free Survival (PFS) Rate at 3 Months Based on Independent Central Review (ICR)
Description: as for outcome 3
Time Frame: Tumour assessments every 6 weeks from 1st dose of treatment until Recist 1.1 defined radiological progressive disease. Calculated at 3 months using the Kaplan-Meier technique
Population: HER2-positive Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 73
Percentage of participants | 69.0 [56.8 to 78.4]

5. Secondary Outcome: Progression-free Survival (PFS) Rate at 6 Months Based on Independent Central Review (ICR)
Description: as for outcome 3
Time Frame: Tumour assessments every 6 weeks from 1st dose of treatment until Recist 1.1 defined radiological progressive disease. Calculated at 6 months using the Kaplan-Meier technique
Population: HER2-positive Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 73
Percentage of participants | 43.4 [30.8 to 55.3]

6. Secondary Outcome: Progression-free Survival (PFS) Rate at 9 Months Based on Independent Central Review (ICR)
Description: as for outcome 3
Time Frame: Tumour assessments every 6 weeks from 1st dose of treatment until Recist 1.1 defined radiological progressive disease. Calculated at 9 months using the Kaplan-Meier technique
Population: HER2-positive Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 73
Percentage of participants | 27.1 [16.2 to 39.3]

7. Secondary Outcome: Progression-free Survival (PFS) Rate at 12 Months Based on Independent Central Review (ICR)
Description: as for outcome 3
Time Frame: Tumour assessments every 6 weeks from 1st dose of treatment until Recist 1.1 defined radiological progressive disease. Calculated at 12 months using the Kaplan-Meier technique
Population: HER2-positive Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 73
Percentage of participants | 16.7 [8.0 to 28.1]

8. Secondary Outcome: Progression-free Survival (PFS) Rate at 15 Months Based on Independent Central Review (ICR)
Description: as for outcome 3
Time Frame: Tumour assessments every 6 weeks from 1st dose of treatment until Recist 1.1 defined radiological progressive disease. Calculated at 15 months using the Kaplan-Meier technique
Population: HER2-positive Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 73
Percentage of participants | 11.9 [4.7 to 22.8]

9. Secondary Outcome: Progression-free Survival (PFS) Rate at 18 Months Based on Independent Central Review (ICR)
Description: as for outcome 3
Time Frame: Tumour assessments every 6 weeks from 1st dose of treatment until Recist 1.1 defined radiological progressive disease. Calculated at 18 months using the Kaplan-Meier technique
Population: HER2-positive Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 73
Percentage of participants | 4.0 [0.4 to 15.6]

10. Secondary Outcome: Progression-free Survival (PFS) Rate at 21 Months Based on Independent Central Review (ICR)
Description: as for outcome 3
Time Frame: Tumour assessments every 6 weeks from 1st dose of treatment until Recist 1.1 defined radiological progressive disease. Calculated at 21 months using the Kaplan-Meier technique
Population: HER2-positive Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 73
Percentage of participants | 4.0 [0.4 to 15.6]

11. Secondary Outcome: Disease Control Rate (DCR) Based on Independent Central Review (ICR)
Description: Disease control rate based on ICR according to RECIST version 1.1 was defined as the rate of best objective response of complete response (CR), partial response (PR) or stable disease (SD)
Time Frame: as for outcome 3
Population: HER2-positive Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 73
Percentage of participants | 79.5 [68.4 to 88.0]

12. Secondary Outcome: Disease Control Rate (DCR) Based on Independent Central Review (ICR) at Week 12
Description: Disease control rate based on ICR according to RECIST version 1.1 was defined as the rate of best objective response of complete response (CR), partial response (PR) or stable disease (SD) for at least 11 weeks (ie 12 weeks - 1 week to allow for an early assessment within the assessment window)
Time Frame: Tumour assessments every 6 weeks from 1st dose of treatment until Recist 1.1 defined radiological progressive disease. DCR assessed at Week 12
Population: HER2-positive Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 73
Percentage of participants | 74.0 [62.4 to 83.5]

13. Secondary Outcome: Duration of Response (DoR) Based on Independent Central Review (ICR)
Description: DoR defined as the time from the date of first documented OR (confirmed CR or confirmed PR) until date of documented progression (PD) or death in the absence of progression based on investigator assessments by using RECIST version 1.1
Time Frame: as for outcome 3
Population: HER2-positive Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 73
Months | 6.7 [4.6 to 8.8]

14. Secondary Outcome: Overall Survival (OS) Based on Independent Central Review (ICR)
Description: OS based on ICR is defined as the time from date of enrolment until the date of death due to any cause
Time Frame: From date of enrolment until death due to any cause. Assessed up to approximately 30 months (from date of first subject in to data cut-off 28February2024)
Population: HER2-positive Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 73
Months | 11.1 [7.7 to 13.7]

15. Secondary Outcome: Best Percentage Change in Sum of Diameters of Measurable Tumours Based on Independent Central Review (ICR)
Description: Best percentage change based on ICR is defined as the best change in target lesion tumour size from baseline (maximum reduction or minimum increase from baseline in the absence of a reduction)
Time Frame: as for outcome 3
Population: HER2-positive Full analysis set
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 73
Percentage Change | -22.55 (29.682)

ADVERSE EVENTS:
Time Frame: From the signature of the informed consent form until 40 (+7) days after the last dose of study treatment or until the start of the first subsequent anticancer therapy after discontinuation of study treatment, whichever comes first (maximum treatment duration of 19.3 months)
Groups:
- T-DXd: Description (Arm-group)
Arm/Group | T-DXd
All-Cause Mortality (participants affected / at risk) | 77/95
Serious Adverse Events (participants affected / at risk) | 40/95
Other Adverse Events (participants affected / at risk) | 93/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T-DXd (N=95)
Dysphagia (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 5
Hepatic function abnormal (Hepatobiliary disorders) | 2
Jaundice cholestatic (Hepatobiliary disorders) | 1
Covid-19 pneumonia (Infections and infestations) | 4
Gastrointestinal infection (Infections and infestations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Myelosuppression (Blood and lymphatic system disorders) | 1
Platelet count decreased (Investigations) | 6
White blood cell count decreased (Investigations) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Malnutrition (Metabolism and nutrition disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Death (General disorders) | 2
Fatigue (General disorders) | 1
Covid-19 (Infections and infestations) | 5
Pneumonia (Infections and infestations) | 5
Sepsis (Infections and infestations) | 1
Neutrophil count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Haemorrhage intracranial (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T-DXd (N=95)
Diarrhoea (Gastrointestinal disorders) | 14
Nausea (Gastrointestinal disorders) | 41
Asthenia (General disorders) | 24
Anaemia (Blood and lymphatic system disorders) | 73
Fatigue (General disorders) | 18
Oedema peripheral (General disorders) | 7
Hepatic function abnormal (Hepatobiliary disorders) | 5
Covid-19 (Infections and infestations) | 12
Alanine aminotransferase increased (Investigations) | 24
Amylase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 30
Bilirubin conjugated increased (Investigations) | 6
Blood alkaline phosphatase increased (Investigations) | 11
Blood bilirubin increased (Investigations) | 11
Blood creatinine increased (Investigations) | 6
Blood lactate dehydrogenase increased (Investigations) | 5
Ejection fraction decreased (Investigations) | 5
Gamma-glutamyltransferase increased (Investigations) | 11
Lymphocyte count decreased (Investigations) | 16
Neutrophil count decreased (Investigations) | 58
Platelet count decreased (Investigations) | 50
Weight decreased (Investigations) | 27
White blood cell count decreased (Investigations) | 69
White blood cell count increased (Investigations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 38
Hyperglycaemia (Metabolism and nutrition disorders) | 8
Hyperuricaemia (Metabolism and nutrition disorders) | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 37
Hypocalcaemia (Metabolism and nutrition disorders) | 23
Hypochloraemia (Metabolism and nutrition disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 25
Hypoproteinaemia (Metabolism and nutrition disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Abdominal distension (Gastrointestinal disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 18
Dyspepsia (Gastrointestinal disorders) | 6
Mouth ulceration (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 30
Pyrexia (General disorders) | 9
Coronavirus infection (Infections and infestations) | 5
Hyponatraemia (Metabolism and nutrition disorders) | 21
Hypoaesthesia (Nervous system disorders) | 6
Insomnia (Psychiatric disorders) | 7
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT04989816/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT04989816/SAP_001.pdf